CLINICAL TRIAL: NCT01828775
Title: Integration of Palliative Care for Cancer Patients on Phase I Trials
Brief Title: Palliative Care Intervention in Improving Quality of Life, Psychological Distress, and Communication in Patients With Solid Tumors Receiving Treatment
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: City of Hope Medical Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 13193; NCI-2013-00731 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 1R01CA177562-01A1 (NIH)
Record Dates: First submitted 2013-04-02; First posted 2013-04-11 (Estimated); Last update posted 2021-03-10 (Actual); Status verified 2021-03

CONDITIONS: Unspecified Adult Solid Tumor, Protocol Specific
MeSH Terms: interventions — Palliative Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Arm I (early PCI) (Experimental): Patients receive part I of the PCI comprising quantitative surveys, comprehensive palliative care assessment by the Research Nurses, and goals of care discussions beginning prior to administration of the first dose of phase I treatment. Patients then receive part II of the PCI comprising recommendations from the interdisciplinary team, patient educational sessions, and supportive care referrals following the first dose of phase I treatment and is completed within one month of the first treatment.
  Interventions: Other: palliative care; Procedure: quality-of-life assessment; Other: survey administration
- Arm II (delayed PCI) (Experimental): Patients receive usual care until 12 weeks post-treatment initiation. Patients then receive both part I and II of the PCI.
  Interventions: Other: palliative care; Procedure: quality-of-life assessment; Other: survey administration

INTERVENTIONS:
Other: palliative care — Receive early PCI
  Arms: Arm I (early PCI)
Other: palliative care — Receive delayed PCI
  Arms: Arm II (delayed PCI)
Procedure: quality-of-life assessment — Ancillary studies
  Other Names: quality of life assessment
Other: survey administration — Ancillary studies

SUMMARY:
This pilot randomized clinical trial studies palliative care intervention in improving quality of life, psychological distress, and communication in patients with solid tumors receiving treatment on phase I trials. Cancer patients experience many symptoms related to treatment and the cancer itself that can be distressing and impact quality of life. Palliative care focuses on managing these symptoms and may help patients with solid tumors live more comfortably.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Test the effects of a palliative care intervention (PCI) on patients' quality of life (QOL), psychological distress and satisfaction with communication, comparing the experimental versus control groups.

II. Test the effects of a PCI on patients' symptom intensity and symptom interference with daily activities, comparing the experimental versus control groups.

III. Test the effects of a PCI on patients' hospital and palliative care resource utilization and clinical trial retention rates, comparing the experimental versus control groups.

IV. Test the effects of the timing of PCI initiation (early versus delayed) on patient outcomes, comparing the experimental versus control groups.

V. Describe patients' satisfaction with the PCI.

OUTLINE: Patients are randomized to 1 of 2 arms.

ARM I: Patients receive part I of the PCI comprising quantitative surveys, comprehensive palliative care assessment by the Research Nurses, and goals of care discussions beginning prior to administration of the first dose of phase I treatment. Patients then receive part II of the PCI comprising recommendations from the interdisciplinary team, patient educational sessions, and supportive care referrals following the first dose of phase I treatment and is completed within one month of the first treatment.

ARM II: Patients receive usual care until 12 weeks post-treatment initiation. Patients then receive both part I and II of the PCI.

After completion of study, patients are followed up for 5 years.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with solid tumors who are eligible for participation in Phase I clinical trials of investigational cancer therapies
* Patients who have signed an informed consent for participation in Phase I clinical trials
* Able to read or understand English-this is included because the intervention and study materials (including outcome measures) are only in English
* Ability to read and/or understand the study protocol requirements, and provide written informed consent

Exclusion Criteria:

* Patients diagnosed with hematologic (as a population distinct from solid tumors and different trials) cancers.

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 480 (Actual)
Dates: Start 2014-09-08 (Actual); Primary Completion 2020-05-18 (Actual); Study Completion 2020-05-18 (Actual)

PRIMARY OUTCOMES:
Change in overall QOL scores, assessed by the Functional Assessment of Cancer Therapy-General (FACT-G) and Functional Assessment of Chronic Illness Therapy-Spirituality (FACIT-Sp) | Baseline to 12 weeks
  To control for inflation of experimentwise error caused by analyzing four different QOL subscales, alpha will be set to .01. A 2x2 multiply repeated measures ANCOVA (in which the within groups variables are QOL subscale scores at 4 and 12 weeks, the between groups measure is treatment group (control vs. PCI), and the covariate is baseline QOL) might be employed if the correlation between the four FACT-G subscale scores are high enough to warrant such an analysis. The overall QOL score derived from the FACT-G will be tested individually using alpha=.05.
  If subscale correlations are not high, outcome will be analyzed using four 2x2 repeated measures ANCOVAs in which the within groups variable is each QOL subscale, the between groups measure is group (PCI vs. control), and the covariate is the appropriate baseline QOL subscale (Physical well-being, emotional well-being, social well-being, and functional well-being).
Change in psychological distress, assessed using the Psychological Distress Thermometer | Baseline to 12 weeks
  Analyzed using a 2x2 repeated measures ANCOVA to test for differences in psychological distress (Psychological Distress Thermometer scores), at 4 and 12-week between the PCI and control groups, controlling for baseline psychological distress.
Satisfaction with communication, measured by the Family Satisfaction with Advanced Cancer Care (FAMCARE) | 12 weeks
  Analyzed using a 2x2 repeated measures ANCOVA to test for differences in satisfaction (Family Satisfaction with Advanced Cancer Care scores), at 4 and 12-week between the PCI and control groups, controlling for baseline satisfaction.
Patients' symptom intensity and symptom interference with daily activities | 12 weeks
  Analyzed using a 2x2 repeated measures ANCOVA to test for differences in symptom intensity and symptom interference with daily activities (using Psychological Patient-Reported Outcomes Version of the Common Terminology Criteria for Adverse Events (PRO - CTCAE) scores), at 4 and 12-week between the PCI and control groups, controlling for baseline symptom intensity and symptom interference.
Total numbers of supportive care referrals (social work, dietitian, chaplaincy, psychologist/psychiatrist) | 12 weeks
  Contingency table analysis and the chi square statistic will be used to examine the association between group and referral to various support services. In addition, total number of referrals will be counted and an independent student's t-test will be used to test for significant differences in number of total referrals between groups.
Total number of unscheduled outpatient encounters and inpatient admissions | 12 weeks
  Total number of encounters and admissions will be counted and an independent student's t-test for each variable will be used to test for significant differences in number of total encounters and number of unscheduled admissions between groups.
Total number of hospice referrals | 12 weeks
  Contingency table analysis with the chi square statistic to examine the association between group and hospice referral.
Retention on the Phase I trial | 12 weeks
  Contingency table analysis with the chi square statistic to examine the association between group and Phase I trial retention.
Patient satisfaction with the PCI | 12 weeks
  Descriptive statistics and comparisons between the two groups will be conducted for overall satisfaction with intervention content and timing of the intervention.

SECONDARY OUTCOMES:
Change in overall QOL scores, assessed by FACT-G and FACIT-Sp | Baseline to 4 weeks
  To control for inflation of experimentwise error caused by analyzing four different QOL subscales, alpha will be set to .01. A 2x2 multiply repeated measures ANCOVA (in which the within groups variables are QOL subscale scores at 4 weeks, the between groups measure is treatment group (control vs. PCI), and the covariate is baseline QOL) might be employed if the correlation between the four FACT-G subscale scores are high enough to warrant such an analysis. The overall QOL score derived from the FACT-G will be tested individually using alpha=.05.
  If subscale correlations are not high, outcome will be analyzed using four 2x2 repeated measures ANCOVAs in which the within groups variable is each QOL subscale, the between groups measure is group (PCI vs. control), and the covariate is the appropriate baseline QOL subscale (Physical well-being, emotional well-being, social well-being, and functional well-being).
Change in overall QOL scores, assessed by FACT-G and FACIT-Sp | Baseline to 24 weeks
  To control for inflation of experimentwise error caused by analyzing four different QOL subscales, alpha will be set to .01. A 2x2 multiply repeated measures ANCOVA (in which the within groups variables are QOL subscale scores at 24 weeks, the between groups measure is treatment group (control vs. PCI), and the covariate is baseline QOL) might be employed if the correlation between the four FACT-G subscale scores are high enough to warrant such an analysis. The overall QOL score derived from the FACT-G will be tested individually using alpha=.05.
  If subscale correlations are not high, outcome will be analyzed using four 2x2 repeated measures ANCOVAs in which the within groups variable is each QOL subscale, the between groups measure is group (PCI vs. control), and the covariate is the appropriate baseline QOL subscale (Physical well-being, emotional well-being, social well-being, and functional well-being).
Change in psychological distress, assessed using the Psychological Distress Thermometer | Baseline to 4 weeks
  Analyzed using a 2x2 repeated measures ANCOVA to test for differences in psychological distress (Psychological Distress Thermometer scores), at 4 weeks, between the PCI and control groups, controlling for baseline psychological distress.
Change in psychological distress, assessed using the Psychological Distress Thermometer | Baseline to 24 weeks
  Analyzed using a 2x2 repeated measures ANCOVA to test for differences in psychological distress (Psychological Distress Thermometer scores), at 24 weeks, between the PCI and control groups, controlling for baseline psychological distress.
Satisfaction with communication, measured by FAMCARE | 4 weeks
  Analyzed using a 2x2 repeated measures ANCOVA to test for differences in satisfaction (Family Satisfaction with Advanced Cancer Care scores), at 4 weeks, between the PCI and control groups, controlling for baseline satisfaction.
Satisfaction with communication, measured by FAMCARE | Up to 24 weeks
  Analyzed using a 2x2 repeated measures ANCOVA to test for differences in satisfaction (Family Satisfaction with Advanced Cancer Care scores), up to 24 weeks, between the PCI and control groups, controlling for baseline satisfaction.
Patients' symptom intensity and symptom interference with daily activities | Up to 24 weeks
  Analyzed using a 2x2 repeated measures ANCOVA to test for differences in symptom intensity and symptom interference with daily activities (Patient-Reported Outcomes Version of the Common Terminology Criteria for Adverse Events (PRO - CTCAE) scores), up to 24 weeks, between the PCI and control groups, controlling for baseline satisfaction.
Total numbers of supportive care referrals (social work, dietitian, chaplaincy, psychologist/psychiatrist) | Up to 24 weeks
  Contingency table analysis and the chi square statistic will be used to examine the association between group and referral to various support services for up to 24 weeks. In addition, total number of referrals will be counted and an independent student's t-test will be used to test for significant differences in number of total referrals between groups.
Total number of unscheduled outpatient encounters and inpatient admissions | Up to 24 weeks
  Total number of encounters and admissions will be counted and an independent student's t-test for each variable will be used to test for significant differences in number of total encounters and number of unscheduled admissions between groups for up to 24 weeks.
Total number of hospice referrals | Up to 24 weeks
  Contingency table analysis with the chi square statistic to examine the association between group and hospice referral for up to 24 weeks.
Retention on the Phase I trial | Up to 24 weeks
  Contingency table analysis with the chi square statistic to examine the association between group and Phase I trial retention for up to 24 weeks.
Patient satisfaction with the PCI | Up to 24 weeks
  Descriptive statistics and comparisons between the two groups will be conducted for overall satisfaction with intervention content and timing of the intervention for up to 24 weeks.

CONTACTS AND LOCATIONS:
Overall Officials: Betty Ferrell, Principal Investigator — City of Hope Medical Center
Locations (2):
- United States (2):
  - City of Hope Medical Center, Duarte, California
  - Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins Hospital, Baltimore, Maryland